CLINICAL TRIAL: NCT06425809
Title: Predictors of Muscle Injury Risk in Non-professional Football Players From the Principality of Asturias. An Ambispective Cohort Study.
Brief Title: Predictors of Muscle Injury Risk in Non-professional Football Players
Status: Completed | Type: Observational
Sponsor: University of Oviedo (Other)
Responsible Party: Principal Investigator, Ruben Cuesta Barriuso, Principal Investigator, University of Oviedo
Other Study IDs: Pred-Fut
Record Dates: First submitted 2024-05-14; First posted 2024-05-22 (Actual); Last update posted 2025-03-26 (Actual); Status verified 2024-05

CONDITIONS: Sport Injury
Keywords: Muscular Diseases; Football; Risk; Secondary Prevention; Physiotherapy
MeSH Terms: conditions — Muscular Diseases | interventions — Observation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Observational group: Data collection will take place between May and June 2024. This will be done through a self-questionnaire format with closed questions where no data will be collected that allow the identification of the subject (name, surname, or national identity document).
  The coding of the data collected and its analysis will be carried out under the supervision of the principal investigator, in accordance with current data protection regulations, scrupulously complying with the anonymous collection of clinical data, and without collecting any data that could allow the identification of the patients whose data are collected.
  Interventions: Other: Observation

INTERVENTIONS:
Other: Observation — The data collection will be carried out by the two researchers, in accordance with current data protection regulations, scrupulously complying with the anonymous collection of clinical data, and without collecting any data that could allow the identification of the athletes whose data are collected. The members of the research group will not have access to personal data that could facilitate the identity of any person on the basis of the data collected. The data collected in this study, anonymised from the outset, will be exported to an Excel file. Access to the Excel file will require password access and will be managed from a computer of the University of Oviedo (Department of Surgery and Medical-Surgical Specialities).

SUMMARY:
Background. Football accounts for 30% of all sports injuries. Muscle injuries in football are the most common non-traumatic and non-contact injuries. A comprehensive approach to injury prevention must consider the design of the footwear and the environmental conditions in which the match is played.

Objective. To assess the risk of injury as a function of footwear and field of play in non-professional football players and to identify the best predictive model of muscle injury in these athletes.

Method. Ambispective cohort study. Ninety-seven players will be recruited. The primary variable will be the number of lower limb muscle injuries in the last 3 seasons. Secondary and modifying variables will be: age, body mass index, boot type, pitch turf, training load and field position. Potential confounding variables will be motivation for choice of footwear, date of muscle injuries, time playing in the category and presence in the starting team. The analysis will calculate the risk of adverse effects in these patients and assess the influence of confounders and trend analysis on the primary variable, stratified by potential confounders.

Expected outcomes. To calculate the risk of muscle injury as a function of anthropometric variables, and footwear and turf type. To identify the predictive model of muscle injuries in football players.

ELIGIBILITY:
Inclusion Criteria:

* Federated, non-professional football players.
* Competing in category 3 RFEF (group 2).
* Who compete in the territorial delimitation of the Principality of Asturias.
* Subjects who have not undergone previous musculoskeletal surgery in the seasons under study.
* Who were federated at least one year before the study period.

Exclusion Criteria:

* Players who have not participated in competition, during the seasons under study, for a period of more than 6 months due to a musculoskeletal injury.

Ages: 18 Years to 30 Years | Sex: Male
Age Groups: Adult
Study Population: Population: Non-professional football players from the Principality of Asturias, where the aim is to identify the risk of muscle injuries in these players and to identify the predictive model of muscle injuries based on anthropometric and sporting variables.
Sampling Method: Non-Probability Sample
Enrollment: 156 (Actual)
Dates: Start 2024-05-20 (Actual); Primary Completion 2024-06-15 (Actual); Study Completion 2024-07-01 (Actual)

PRIMARY OUTCOMES:
Asses the number of lower limb muscle injuries in the last 3 competition seasons | Screening visit
  The primary variable, the number of lower limb muscle injuries in the last 3 seasons, will be assessed as a quantitative variable.

SECONDARY OUTCOMES:
Assess the age | Screening visit
  The secondary variable, age (in years completed), will be assessed as a quantitative variable.
Assess the body mass index | Screening visit
  The secondary variable, body mass index (in kg/m2), will be assessed as a quantitative variable.
Assess the type of training and competition boot in the last 3 competition seasons | Screening visit
  The secondary variable, type of training and competition boot (rubber cleat/metal cleat), will be assessed as a nominal qualitative variable.
Assess the type of training and competition pitch in the last 3 competition seasons | Screening visit
  The secondary variable, type of training and competition pitch (sand pitch / artificial turf pitch / natural grass pitch), will be assessed as a nominal qualitative variable.
Assess the type of muscle injury in the last 3 competition seasons | Screening visit
  The secondary variable, type of muscle injury (fibrillar / musculotendinous / strain), will be assessed as an ordinal qualitative variable.
Assess the weekly training load in the last 3 competition seasons | Screening visit
  The secondary variable, weekly training load (hours/week), will be assessed as a quantitative variable.
Assess the position on the field in the last 3 competition seasons | Screening visit
  The secondary variable, position on the field (goalkeeper / defender / midfielder / striker), will be assessed as an ordinal qualitative variable.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Oviedo, Oviedo, Principality of Asturias, Spain